CLINICAL TRIAL: NCT06409689
Title: Enhanced Postoperative Analgesia and Accelerated Recovery With Oliceridine: A Study on G-Protein Biased μ-Opioid Agonist
Brief Title: Oliceridine-Enhanced Analgesia and Recovery: A G-Protein Biased μ-Opioid Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Hui Xu, professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S058
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Analgesia
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oliceridine fumarate low dose group (Experimental): The first loading dose of oliceridine fumarate was 1.5 mg in all patients after operation. The PCA dose of the patients was 0.1 mg, and the locking interval was 6 min. A supplemental dose of 0.75 mg is allowed once per hour as needed after 1 h of the load dose; The maximum cumulative daily dose is 27mg. The duration of PCA analgesia was 48 hours.
  Interventions: Drug: Oliceridine fumarate low dose
- Oliceridine fumarate medium dose group (Experimental): The first loading dose of oliceridine fumarate was 1.5 mg in all patients after operation. The PCA dose of the patients was 0.35mg, and the locking interval was 6 min. A supplemental dose of 0.75 mg is allowed once per hour as needed after 1 h of the load dose; The maximum cumulative daily dose is 27mg. The duration of PCA analgesia was 48 hours.
  Interventions: Drug: Oliceridine fumarate moderate dose
- Oliceridine fumarate high dose group (Experimental): The first loading dose of oliceridine fumarate was 1.5 mg in all patients after operation. The PCA dose of the patients was 0.5 mg, and the locking interval was 6 min. A supplemental dose of 0.75 mg is allowed once per hour as needed after 1 h of the load dose; The maximum cumulative daily dose is 27mg. The duration of PCA analgesia was 48 hours.
  Interventions: Drug: Oliceridine fumarate high dose
- Morphine group (Experimental): The first loading dose of morphine was 4 mg in all patients after operation. The PCA dose of the patients was 1 mg, and the locking interval was 6 min. A supplemental dose of 2 mg is allowed once per hour as needed after 1 h of the load dose; The maximum cumulative daily dose is 60 mg. The duration of PCA analgesia was 48 hours.
  Interventions: Drug: morphine

INTERVENTIONS:
Drug: Oliceridine fumarate low dose — The first loading dose of oliceridine fumarate was 1.5 mg in all patients after operation. The PCA dose of the patients was 0.1 mg, and the locking interval was 6 min. A supplemental dose of 0.75 mg is allowed once per hour as needed after 1 h of the load dose
  Arms: Oliceridine fumarate low dose group
Drug: Oliceridine fumarate high dose — The first loading dose of oliceridine fumarate was 1.5 mg in all patients after operation. The PCA dose of the patients was 0.5 mg, and the locking interval was 6 min. A supplemental dose of 0.75 mg is allowed once per hour as needed after 1 h of the load dose
  Arms: Oliceridine fumarate high dose group
Drug: Oliceridine fumarate moderate dose — The first loading dose of oliceridine fumarate was 1.5 mg in all patients after operation. The PCA dose of the patients was 0.35 mg, and the locking interval was 6 min. A supplemental dose of 0.75 mg is allowed once per hour as needed after 1 h of the load dose
  Arms: Oliceridine fumarate medium dose group
Drug: morphine — The first loading dose of morphine was 4 mg in all patients after operation. The PCA dose of the patients was 1 mg, and the locking interval was 6 min. A supplemental dose of 2 mg is allowed once per hour as needed after 1 h of the load dose; The maximum cumulative daily dose is 60 mg.
  Arms: Morphine group

SUMMARY:
Identifying the lowest effective opioid dose that achieves rapid pain relief while minimizing side effects is a principal objective in postoperative multimodal analgesia strategies. This study aims to determine the optimal analgesic regimen and dosage by assessing the clinical efficacy of oliceridine for postoperative pain management. It also evaluates oliceridine's contribution to accelerated postoperative recovery, examining aspects such as postoperative pulmonary complications, gastrointestinal function, nausea and vomiting, cognitive function, and emotional distress. Furthermore, the study integrates microbiomics and metabolomics to investigate the underlying molecular mechanisms by which oliceridine promotes rapid postoperative recovery. This research will broaden the clinical data and potential applications of oliceridine, addressing gaps in the field and enhancing practical knowledge. Moreover, this is the first time a clinical study combining multiple omics approaches will provide a comprehensive theoretical foundation for its clinical benefits.

DETAILED DESCRIPTION:
This study selects 80 elective patients slated for upper abdominal laparoscopic surgery under general anesthesia, classified as ASA I-II. These patients are randomly allocated into four groups: Oliceridine low dose (OⅠ), medium dose (OⅡ), and high dose (OⅢ), and a Morphine (M) group. The postoperative analgesic protocol includes a universal loading dose of 1.5 mg for all groups. Depending on the group, the PCA doses are set at 0.1 mg, 0.35 mg, or 0.5 mg, with a lockout interval of 6 minutes. After the initial dose, patients may receive an additional 0.75 mg per hour as needed, with a daily ceiling of 27 mg for Oliceridine. In the Morphine group, the loading dose is 4 mg with a PCA dose of 1 mg and similar lockout, allowing 2 mg per hour post-loading, capped at 60 mg daily. Outcomes to monitor include systolic and diastolic blood pressures, heart rate, oxygen saturation, and respiratory rate at 6, 24, and 48 hours postoperatively; pain levels using the NRS scale; nausea and vomiting via the VAS score; and pulmonary complications evaluated by EPCO standards at specified intervals. Gastrointestinal function is assessed using the I-FEED score, and mental health through the HADS scale preoperatively and 48 hours post-surgery. Cognitive function is evaluated using the MMSE scale preoperatively and 72 hours postoperatively. Patient fecal samples are collected pre- and 48 hours post-surgery for microbial and metabolomic analyses to identify potential molecular benefits of Oliceridine, informed by its G-protein biased pharmacology. The study also uses statistical methods to compare microbiological outcomes and correlate these with clinical presentations.

ELIGIBILITY:
Inclusion Criteria:

1. ASA grades 1-2
2. Age > 18 years and < 70 years
3. Laparoscopic upper abdominal surgery under general anesthesia is planned, and the operation time is not more than 4 hours
4. Voluntarily receive postoperative controlled intravenous analgesia
5. Subjects understand and can cooperate with this study
6. Subjects can provide and sign written informed consent prior to conducting investigation-related screening procedures

Exclusion Criteria:

1. BMI>30 kg/m2 or < 19 kg/m2
2. Patients with preoperative use of opioids, acute and chronic pain or hyperalgesia
3. Patients with coronary atherosclerotic heart disease, significant ischemic heart disease, severe angina, heart failure, valvular disease or other heart disease
4. More severe hepatic and renal insufficiency
5. A history of mental illness or alcoholism
6. A history of alcohol or drug abuse
7. Combined with cranial pressure, intraocular pressure or glaucoma
8. Poorly controlled or untreated hypertension before surgery
9. Preeclampsia or eclampsia
10. Untreated and undertreated hyperthyroidism
11. Combined with autoimmune disease
12. Unable to use the numerical rating scale
13. History of chronic cough
14. Surgery is expected to take more than 4 hours Patients enrolled in other clinical trials within 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain score | 6 hour, 24hour, and 48 hour after surgery
  The NRS Numerical Pain Evaluation Scale assessed postoperative pain status: no pain (0), mild pain (1-3), moderate pain (4-6), and severe pain (7-10).

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | 6 hour, 24 hour, and 48 hour after surgery
  With a 10cm ruler as the scale, 0 at one end indicates no nausea and vomiting, and 10 at the other end indicates the most severe nausea and vomiting that is unbearable. 1 to 4 is mild, 5 to 6 is moderate, 7 to 10 is severe
Postoperative pulmonary complications | 24 hour,72 hour after surgery
  european perioperative clinical outcome (EPCO)
Postoperative cognitive function | Before surgery, 3 days after surgery
  (mini-mental state examination, MMSE) scale score，The maximum score is 30 points. The classification of dementia is related to the level of education, so if the elderly are illiterate and less than 17 points, primary school and less than 20 points, secondary school and above less than 24 points, then dementia.
Flora abundance | One day before surgery and 48 hours after surgery
  Feces were collected from patients before surgery and 48 hours after surgery (stored at negative 80 degrees), and the fecal intestinal flora abundance of patients in each group was determined by 16S rRNA omics

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China